CLINICAL TRIAL: NCT01430260
Title: A Multi-center, Open, Randomized, Three-arm, Parallel-group, Phase IV Study to Compare the Efficacy of Ciclesonide Nasal Spray and Levocetirizine, Alone and in Combination for the Patient With Allergic Rhinitis
Brief Title: Omnaris Versus Levocetirizine Phase 4 Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HANDOK2010.07
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-09

CONDITIONS: Allergic Rhinitis
Keywords: efficacy; ciclesonide; levocetirizine; allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — ciclesonide; levocetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ciclesonide nasal spray (Experimental): ciclesonide nasal spray, alone
  Interventions: Drug: Ciclesonide
- Levocetirizine (Active Comparator): Levocetirizine, alone
  Interventions: Drug: Levocetirizine
- Ciclesonide nasal spray & Levocetirizine (Active Comparator): Ciclesonide nasal spray & Levocetirizine in combination
  Interventions: Drug: Ciclesonide & Levocetirizine

INTERVENTIONS:
Drug: Ciclesonide — 200 ㎍ once daily
  Other Names: Omnaris
  Arms: ciclesonide nasal spray
Drug: Levocetirizine — 5mg once daily
  Other Names: XYZAL
  Arms: Levocetirizine
Drug: Ciclesonide & Levocetirizine — * Omnaris (ciclesonide) 200 ㎍ once daily
  * Levocetirizine 5mg once daily
  Other Names: Omnaris nasal spray; XYZAL
  Arms: Ciclesonide nasal spray & Levocetirizine

SUMMARY:
This i a comparison of the efficacy ciclesonide nasal spray and levocetirizine, alone and in combination.

DETAILED DESCRIPTION:
randomized, open-label, three arm, parallel group, multi-center study

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinitis patients aged ≥ 18 years (with a history of AR of 1 years or longer)
* Moderate to severe patient according to ARIA guideline
* To have a demonstrated positive skin prick test or other serologic tests to at least 1 allergen.
* Subjects who complete the subject diary(S) at least 70%.

Exclusion Criteria:

* Nasal pathology, including nasal polyps, clinically relevant respiratory tract malformations, recent nasal biopsy (within 60 days), nasal trauma, nasal surgery, atrophic rhinitis, rhinitis medicamentosa (within 60 days), asthma requiring corticosteroid treatment
* Hypersensitivity to corticosteroid and/or hydroxyzine
* Hypersensitivity to galactose intolerance, lapp lactase deficiency, glucose-galactose malabsorption
* A history of respiratory tract infection or disorder within 2 weeks of the screening visit or had a respiratory tract infection during baseline
* Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of β-agonists
* Treated with systemic corticosteroids (within 8 weeks of study initiation) or topical corticosteroids (> 1% hydrocortisone, within 4 weeks of study initiation) or antibiotics (within 2 weeks of first visit)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
rTNSS | 2 weeks
  change from baseline in the average of AM and PM patient assessed reflective TNSS

SECONDARY OUTCOMES:
rTOSS | 2 weeks
  Reflective total ocular symptom sores
TNSS | 2 weeks
  Patient assessed individual TNSS
PANS | 2 weeks
  Physician-assessed overall nasal signs and symptoms severity (PANS)
RQLQ | 2 weeks
  Rhinoconjunctivitis quality of life questionnaire (RQLQ)

CONTACTS AND LOCATIONS:
Overall Officials: Moonhwa Park, Doctor, Study Director — Handok Inc.
Locations (1):
- handok pharmaceuticals co. LTD, Seoul, Seoul, South Korea